CLINICAL TRIAL: NCT00317395
Title: A Randomized, Double-blind, Triple-dummy, Dose-ranging Study, Including an Active Control of Unfractionated Heparin and Eptifibatide, to Evaluate the Clinical Efficacy and Safety of Otamixaban, in Patients With Non-ST Elevation Acute Coronary Syndrome and Planned Early Invasive Strategy
Brief Title: Study of Otamixaban Versus Unfractionated Heparin (UFH) and Eptifibatide in Non-ST Elevation Acute Coronary Syndrome
Acronym: SEPIA-ACS1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6624; XRP0673A/2003 (Other: HMR); 2006-000506-22 (EudraCT Number)
Record Dates: First submitted 2006-04-21; First posted 2006-04-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Coronary Disease
Keywords: Non ST elevation Acute Coronary Syndrome; Early invasive strategy; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Disease | interventions — otamixaban; Heparin; Eptifibatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Otamixaban Dose 1 (Experimental): dosage regimen 1
  Interventions: Drug: Otamixaban (XRP0673)
- Otamixaban Dose 2 (Experimental): dosage regimen 2
  Interventions: Drug: Otamixaban (XRP0673)
- Otamixaban Dose 3 (Experimental): dosage regimen 3
  Interventions: Drug: Otamixaban (XRP0673)
- Otamixaban Dose 4 (Experimental): dosage regimen 4
  Interventions: Drug: Otamixaban (XRP0673)
- Otamixaban Dose 5 (Experimental): dosage regimen 5
  Interventions: Drug: Otamixaban (XRP0673)
- UFH/Eptifibatide (Active Comparator)
  Interventions: Drug: unfractionated heparin; Drug: eptifibatide

INTERVENTIONS:
Drug: Otamixaban (XRP0673) — intravenous administration
  Arms: Otamixaban Dose 1; Otamixaban Dose 2; Otamixaban Dose 3; Otamixaban Dose 4; Otamixaban Dose 5
Drug: unfractionated heparin — intravenous administration
  Arms: UFH/Eptifibatide
Drug: eptifibatide — intravenous administration
  Arms: UFH/Eptifibatide

SUMMARY:
Primary objective: To demonstrate the clinical efficacy of otamixaban (dose effect via 5 intravenous [IV] regimens) in patients with moderate-to-high-risk non-ST elevation acute coronary syndromes (ACS) and planned early invasive strategy.

Secondary objectives: To evaluate safety and assess pharmacokinetics (PK) and pharmacodynamics (PD).

ELIGIBILITY:
Inclusion Criteria:

* Ischemic discomfort at rest ≥ 10 minutes within 24 hours of randomization
* Electrocardiogram (ECG) criteria for non-ST elevation ACS or cardiac enzyme elevation (> upper limit of normal [ULN])
* No ST elevation Myocardial Infarction (STEMI)
* Planned coronary angiography followed when indicated by a Percutaneous Coronary Intervention (PCI) on Day 1 to Day 3

Exclusion Criteria:

* Inability to undergo coronary angiography or PCI by Day 3
* Prior PCI within 30 days
* Acute STEMI
* Cardiogenic shock
* Anticoagulant treatment for > 24 hours prior to randomization
* Prior treatment with fondaparinux since ACS onset
* Requirement for oral anticoagulant (OAC) prior to Day 30
* Creatinine clearance < 30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3241 (Actual)
Dates: Start 2006-06; Primary Completion 2008-10 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Quadruple efficacy composite of all-cause death, new myocardial infarction, severe recurrent ischemia requiring urgent revascularization and in-hospital bailout use of glycoprotein GPIIb/IIIa inhibitor | within 7 days following randomization

SECONDARY OUTCOMES:
Net clinical benefit: composite of the primary efficacy end point and Thrombolysis in Myocardial Infarction (TIMI) significant bleeding | within 7 days and 30 days following randomization
Quadruple efficacy composite of all-cause death, new myocardial infarction, severe recurrent ischemia requiring urgent revascularization and in-hospital bailout use of glycoprotein GPIIb/IIIa inhibitor | within 30 days, 90 days and 180 days following randomization
Incidence of TIMI significant bleeding | within 7 days following randomization
Incidence of all bleedings | within 7 days and 30 days following randomization

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (36):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Quebec, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Cali, Colombia
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Tatari, Estonia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Bangkok, Thailand
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Sabatine MS, Antman EM, Widimsky P, Ebrahim IO, Kiss RG, Saaiman A, Polasek R, Contant CF, McCabe CH, Braunwald E. Otamixaban for the treatment of patients with non-ST-elevation acute coronary syndromes (SEPIA-ACS1 TIMI 42): a randomised, double-blind, active-controlled, phase 2 trial. Lancet. 2009 Sep 5;374(9692):787-95. doi: 10.1016/S0140-6736(09)61454-9. Epub 2009 Aug 28. PMID 19717184